CLINICAL TRIAL: NCT00419328
Title: NGR002: A Modified Phase I Study of NGR-hTNF in Advanced Solid Tumors: Definition of an Optimal Biological Dose
Brief Title: A Modified Phase I Study of NGR-hTNF in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR002; 2004-002194-23 (EudraCT Number)
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2013-01

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors NGR-hTNF
MeSH Terms: interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Arm A (Experimental): Patients were scheduled to receive a 1 hour intravenous (iv) infusion of NGR-hTNF every 3weeks.- The dose of administered NGR-hTNF was: 0.2, 0.4, 0.8, 1.6 μg/m2 (step 1); 3.2, 6.4, 12.8 μg/m2 (step 2); 19.2, 28.8, 43.2 64.8 μg/m2 (step 3); 86.2, 114.6, 152.4 μg/m2 (step 4)
  Interventions: Drug: NGR-hTNF

INTERVENTIONS:
Drug: NGR-hTNF — Drug: NGR-hTNF
  NGR-hTNF was administered every 3 weeks by a 1 hour intravenous iv infusion. NGR-hTNF in PBS was diluted in 0.9% NaCl, containing human serum albumin.
  Step 1:
  * starting dose: 0.2 μg/m2
  * following doses: 0.4, 0.8 and 1.6 μg/m2.
  * number of patients: 4 per dose level
  Step 2:
  * starting dose: 3.2 μg/m2
  * following doses: 6.4 and 12.8 μg/m2
  * number of patients: 3 per dose level
  Step 3:
  * starting dose: 19.2 μg/m2
  * following doses: 28.8, 43.2 and 64.8 μg/m2
  * number of patients: 3 per dose level
  Step 4:
  * starting dose: 86.2 μg/m2
  * following doses: 114.6 and 152.4 μg/m2
  * number of patients: 3 per dose level
  Other Names: iv q3W escalating dose up 1.6 mcg/sqm

SUMMARY:
The main objective of the trial is to explore the safety and biological activity of NGR-hTNF. The safety will be established by clinical and laboratory assessment. The biological activity will be evaluated by DCE-MRI with contrast media.

DETAILED DESCRIPTION:
This is a modified phase I Single arm, open, non randomized trial of NGR-hTNF in advanced solid tumors for the definition of an optimal biological

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with proven advanced solid tumors not amenable to any clinical improvement by current standard treatments. Tumors recognized to be highly vascularized (e.g. renal, colon thyroid and head and neck cancers), will be included.
* ECOG Performance status 0 - 2
* Patients may have had prior therapy providing the following conditions are met:

  * Chemo, radio, hormonal or immunotherapy: wash-out period of 28 days
  * Surgery: wash-out period of 14 days
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:
* Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
* Bilirubin < 1.5 x ULN
* AST and/or ALT < 2.5 x ULN in absence of liver metastases
* AST and/or ALT < 5 x ULN in presence of liver metastases
* Serum creatinine < 1.5 x ULN
* Absence of any conditions in which hypervolemia and its consequences (e.g. increased stroke volume, elevated blood pressure) or haemodilution could represent a risk for the patient (reference appendix "Technical data sheet human albumin")
* Normal cardiac function and absence of uncontrolled hypertension
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients may not receive any other investigational agents while on study
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To verify safety of escalating doses of NGR-hTNF | during and following the treatment
  To verify safety of escalating doses of NGR-hTNF

SECONDARY OUTCOMES:
To document possible modifications on vessels permeability | before and following the first treatment
  To document possible modifications on vessels permeability
To document signs of anticancer activity | every 6 weeks
  To document signs of anticancer activity

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (1):
- Fondazione San Raffaele del Monte Tabor, Milan, Italy

REFERENCES:
- [Result] Gregorc V, Citterio G, Vitali G, Spreafico A, Scifo P, Borri A, Donadoni G, Rossoni G, Corti A, Caligaris-Cappio F, Del Maschio A, Esposito A, De Cobelli F, Dell'Acqua F, Troysi A, Bruzzi P, Lambiase A, Bordignon C. Defining the optimal biological dose of NGR-hTNF, a selective vascular targeting agent, in advanced solid tumours. Eur J Cancer. 2010 Jan;46(1):198-206. doi: 10.1016/j.ejca.2009.10.005. PMID 19900802